CLINICAL TRIAL: NCT03826342
Title: Technology-Based Intervention for Reducing Sexually Transmitted Infections and Substance Use During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Golfo Tzilos, Assistant Professor of Family Medicine and Assistant Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00143896; 1R01HD093611-01A1 (NIH)
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Sexually Transmitted Infection; Alcohol Use Complicating the Puerperium; Alcohol Use Complicating Pregnancy, Unspecified Trimester; Drug Use
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Time

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Check-up for Expectant Moms (Experimental): Theory-driven and derived from empirical support
  Interventions: Behavioral: Health Check-up for Expectant Moms
- Time, attention, and information-matched control (Active Comparator): Well-validated
  Interventions: Behavioral: Time, attention, and information-matched control

INTERVENTIONS:
Behavioral: Health Check-up for Expectant Moms — A brief intervention (one session plus two booster sessions)
  Arms: Health Check-up for Expectant Moms
Behavioral: Time, attention, and information-matched control — We will include facts about alcohol/drug use and risky sex during pregnancy, along with informational brochures that provide face validity.
  Arms: Time, attention, and information-matched control

SUMMARY:
This proposed study is to test whether Health Check-up for Expectant Moms (HCEM), a computer-delivered screening and brief intervention (SBI) that simultaneously targets sexually transmitted infection (STI) risk and alcohol/drug use during pregnancy, reduces antenatal and postpartum risk more than an attention, time, and information matched control condition among pregnant women seeking prenatal care.

ELIGIBILITY:
Inclusion Criteria:

* At least one unprotected vaginal (or anal) sex occasion in the past 30 days
* Having more than one male sex partner in the last 6 months and/or having uncertainty about current partner's monogamy.
* Pregnant
* Current alcohol/drug use risk.

Exclusion Criteria:

* Unable to understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Golfo Tzilos Wernette, Principal Investigator — University of Michigan
Locations (1):
- West Ann Arbor Health Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The study team does not currently have a plan to share data. However, the team is currently in discussion about sharing data and will update the registration as needed.

REFERENCES:
- [Derived] Tzilos Wernette G, Countryman K, Mmeje O, Ngo QM, Zlotnick C. Adapting to the Pandemic: Protocol of a Web-Based Perinatal Health Study to Improve Maternal and Infant Outcomes. JMIR Res Protoc. 2021 Sep 10;10(9):e30367. doi: 10.2196/30367. PMID 34351867

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 180 participants were consented. 4 withdrew from the trial prior to randomization. Since the primary study outcome included measures at the baseline, 2-month follow-up, and 6-month follow-up assessments, a participant was deemed as completing the study if they completed the baseline visit and the 2-month follow-up visit or the 6-month follow-up visit.
Period: Overall Study
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Started | 88 | 88
2 Months | 71 | 76
6 Month | 54 | 59
6 Weeks Post Partum | 68 | 77
Completed | 72 | 77
Not Completed | 16 | 11
Not completed — Withdrawal by Subject | 8 | 1
Not completed — Lost to Follow-up | 7 | 7
Not completed — Miscarriage - Loss of Eligibility to Participate | 1 | 3

BASELINE CHARACTERISTICS:
Population: 180 participants were consented for this trial. 4 withdrew prior to randomization and collection of baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control | Total
Number analyzed (Participants) | 88 | 88 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.26 (4.94) | 30.08 (5.13) | 30.17 (5.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 88 | 176
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 12 | 17
  Not Hispanic or Latino | 83 | 76 | 159
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 27 | 45
  White | 61 | 51 | 112
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88 | 88 | 176

OUTCOME MEASURES:

1. Primary Outcome: Unprotected Sexual Occasions (USOs)
Description: USOs were instances of sexual intercourse where neither partner utilized any form of contraception. Participants were assessed using Timeline Follow-Back (TLFB), a calendar assisted structured interview that provided a way to cue memory so that accurate recall was enhanced for event-level data. TLFB has been used to assess sexual risk-taking. Participants were asked to provide the number of USOs experienced 90 days prior to baseline assessment, between baseline assessment and 2-month follow up, and from 2-month follow up to 6-month follow up.
Time Frame: Up to 6 months
Population: Some participants did not attend the 2-month or 6-month assessments.
Measure: Mean (Standard Deviation); unit: USOs per participant
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Number analyzed (Participants) | 88 | 88
USOs per participant
  Baseline (past 90 days) | 27.73 (37.17) | 41.50 (64.15)
  Baseline to 2-month assessment: number analyzed (Participants) | 71 | 76
  Baseline to 2-month assessment | 8.68 (8.46) | 14.70 (17.61)
  2-month assessment to 6-month assessment: number analyzed (Participants) | 54 | 59
  2-month assessment to 6-month assessment | 11.02 (16.09) | 19.78 (27.89)
Statistical Analysis 1: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; Baseline to 2-month assessment; Test type: Superiority; p = 0.2964, Generalized linear mixed model analysis; generalized linear mixed model analysis under a negative binomial framework
Statistical Analysis 2: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; 2-month assessment to 6-month assessment; Test type: Superiority; p = 0.3404, generalized linear mixed model analysis; generalized linear mixed model analysis under a negative binomial framework

2. Primary Outcome: Alcohol Use Measured by Timeline Follow-Back (TLFB)
Description: Alcohol use was measured by the TLFB. Participants were asked if they had consumed any standard alcoholic drinks 90 days prior to baseline assessment, between baseline assessment and 2-month follow up, and from 2-month follow up to 6-month follow up. Participants' responses could only be Yes or No. Results reflect the participants who responded Yes.
Time Frame: Up to 6 months
Population: Some participants did not attend the 2-month or 6-month assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Number analyzed (Participants) | 88 | 88
Participants
  Baseline (past 90 days) | 61 | 55
  Baseline to 2-month assessment: number analyzed (Participants) | 71 | 76
  Baseline to 2-month assessment | 7 | 5
  2-month to 6-month assessment: number analyzed (Participants) | 54 | 59
  2-month to 6-month assessment | 7 | 2
Statistical Analysis 1: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; Baseline to 2-month assessment; Test type: Superiority; p = 0.7915, Generalized linear mixed model analysis; generalized linear mixed model analysis under a negative binomial framework
Statistical Analysis 2: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; 2-month assessment to 6-month assessment; Test type: Superiority; p = 0.2131, generalized linear mixed model analysis; generalized linear mixed model analysis under a negative binomial framework

3. Primary Outcome: Cannabis Use Measured by Timeline Follow-Back (TLFB)
Description: Cannabis use was measured by the TLFB. Participants were asked if they had used or consumed any cannabis 90 days prior to baseline assessment, between baseline assessment and 2-month follow up, and from 2-month follow up to 6-month follow up. Participants' responses could only be Yes or No. Results reflect the participants who responded Yes.
Time Frame: Up to 6 months
Population: Some participants did not attend the 2-month or 6-month assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Number analyzed (Participants) | 88 | 88
Participants
  Baseline | 25 | 37
  2 month: number analyzed (Participants) | 71 | 76
  2 month | 7 | 12
  6 month: number analyzed (Participants) | 54 | 59
  6 month | 6 | 3
Statistical Analysis 1: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; Baseline to 2-month assessment; Test type: Superiority; p = 0.8357, Generalized linear mixed model analysis; generalized linear mixed model analysis under a negative binomial framework
Statistical Analysis 2: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; 2-month assessment to 6-month assessment; Test type: Superiority; p = 0.0950, generalized linear mixed model analysis; generalized linear mixed model analysis under a negative binomial framework

4. Secondary Outcome: Sexually Transmitted Infections (STIs)
Description: STIs were measured using urine samples or home vaginal swabs testing kits, which were collected at the baseline assessment and 6 weeks postpartum. Results reflect participants whose results came back with positive results for any STI.
Time Frame: Baseline to 6 weeks postpartum (up to 11 months)
Population: Not all participants provided a urine sample or home vaginal swab for testing due to a national shortage on STI tests during the COVID-19 pandemic.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Number analyzed (Participants) | 84 | 78
Participants
  Baseline | 3 | 5
  Up to 6 weeks postpartum: number analyzed (Participants) | 57 | 63
  Up to 6 weeks postpartum | 1 | 3
Statistical Analysis 1: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; Test type: Superiority; p = 0.7496, generalized linear mixed model analysis; generalized linear mixed model analysis under a negative binomial framework

5. Secondary Outcome: Unprotected Sexual Occasions (USOs) Postpartum
Description: USOs were instances of sexual intercourse where neither partner utilized any form of contraception. Participants were assessed using Timeline Follow-Back (TLFB), a calendar assisted structured interview that provided a way to cue memory so that accurate recall was enhanced for event-level data. TLFB has been used to assess sexual risk-taking. Participants were asked to provide the number of USOs experienced from the period of birth up to 6 weeks postpartum.
Time Frame: 6 weeks postpartum (up to 11 months)
Population: Not all participants participated in the postpartum follow-up assessment.
Measure: Mean (Standard Deviation); unit: USOs per participant
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Number analyzed (Participants) | 68 | 77
USOs per participant | 2.24 (7.83) | 2.14 (5.67)
Statistical Analysis 1: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; Test type: Superiority; p = 0.4492, generalized linear mixed model analysis; generalized linear mixed model analysis under a negative binomial framework

6. Secondary Outcome: Birth Weight of Baby
Description: Birth weight of participants' babies was measured in grams.
Time Frame: 6 weeks postpartum (up to 11 months)
Population: Birth weight data was collected from EMRs at the participating sites, regardless of whether the participant completed the 6 Weeks Post Partum visit or not, which is why the Overall Number of Participants Analyzed is different than the Participant Flow. Data from some participants could not be collected because it was missing from the EMR or the participant did not consent to the release of the information. Additionally, data from twins was not included to avoid confounding the results.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Number analyzed (Participants) | 77 | 77
grams | 3412.31 (558.32) | 3244.86 (605.82)
Statistical Analysis 1: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; Test type: Superiority; p = 0.0765, t-test, 2 sided

7. Secondary Outcome: Baby Head Circumference
Description: Head circumference of participants' babies was measured in centimeters.
Time Frame: 6 weeks postpartum (up to 11 months)
Population: Birth head circumference data was collected from EMRs and paper records, regardless of whether the participant completed the 6 Weeks Post Partum visit or not, which is why the Overall Number of Participants Analyzed is different than the Participant Flow. Data from some participants could not be collected because it was missing from the EMR or the participant did not consent to the release of the information. Additionally, data from twins was not included to avoid confounding the results.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Number analyzed (Participants) | 77 | 77
Centimeters | 34.41 (1.80) | 34.20 (2.13)
Statistical Analysis 1: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; Test type: Superiority; p = 0.535, t-test, 2 sided

8. Secondary Outcome: Baby Birth Length
Description: Birth length of participants' babies was measured in centimeters.
Time Frame: 6 weeks postpartum (up to 11 months)
Population: Birth length data was collected from EMRs and paper records, regardless of whether the participant completed the 6 Weeks Post Partum visit or not, which is why the Overall Number of Participants Analyzed is different than the Participant Flow. Data from some participants could not be collected because it was missing from the EMR or the participant did not consent to the release of the information. Additionally, data from twins was not included to avoid confounding the results.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Number analyzed (Participants) | 77 | 77
Centimeters | 50.38 (3.21) | 49.94 (3.51)
Statistical Analysis 1: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; Test type: Superiority; p = 0.4302, t-test, 2 sided

9. Secondary Outcome: Heavy Episodic Drinking
Description: Heavy episodic drinking was defined as consumption of 4 or more standard alcoholic drinks during a single day. Participants were asked if they had engaged in any heavy episodic drinking 90 days prior to baseline assessment and from the period from birth to 6 weeks postpartum. Participants' responses could only be Yes or No. Results reflect the participants who responded Yes.
Time Frame: 6 weeks postpartum (up to 11 months)
Population: Not all participants participated in the postpartum follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Number analyzed (Participants) | 88 | 88
Participants
  Baseline (90 days prior) | 14 | 14
  Birth to 6 weeks postpartum: number analyzed (Participants) | 68 | 77
  Birth to 6 weeks postpartum | 2 | 3
Statistical Analysis 1: Comparison: Health Check-up for Expectant Moms vs Time, Attention, and Information-matched Control; Test type: Superiority; p = 0.8070, generalized linear mixed model analysis; generalized linear mixed model analysis under a negative binomial framework

10. Secondary Outcome: Estimated Cost-effectiveness of Health Check-up for Expectant Moms (HCEM)
Description: Cost-effectiveness was measured in US dollars (USD) and was evaluated as the incremental cost-effectiveness ratio (ICER) that considers the difference in the mean total costs and the difference in health outcomes and events between the two arms. Results reflect the cost-effectiveness evaluation based on estimated costs per case of unprotected sexual occasion averted, alcohol or illicit drug use averted, and sexually transmitted infection (STI) event averted. To develop a plausible full range, a 25% variation of the estimated mean in each arm was used. All participants who were randomized were included in the analysis for this outcome measure.
Time Frame: 6 weeks post-partum (up to 11 months)
Measure: Mean (Full Range); unit: dollars per averted event
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
Number analyzed (Participants) | 88 | 88
dollars per averted event | 3558 [2669 to 4448] | 3380 [2535 to 4225]

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Health Check-up for Expectant Moms | Time, Attention, and Information-matched Control
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/88
Other Adverse Events (participants affected / at risk) | 0/88 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT03826342/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT03826342/ICF_001.pdf